CLINICAL TRIAL: NCT01424449
Title: A Positron Emission Tomography Study in Healthy Male Subjects to Examine the Test-retest Reliability of the D2/3 Agonist Radiotracer [11C]PHNO
Brief Title: A PET Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 113549
Record Dates: First submitted 2011-08-18; First posted 2011-08-29 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-03

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — naxagolide; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no treatment (Experimental): Aripiprazole is a D2/D3 antagonist registered in the UK for use in the treatment of schizophrenia. It allows the highest clinically acceptable blockade of central D2/D3 receptors and will allow us to examine the amount of displaceable binding in the brain - a proposed reference tissue for [11C]PHNO.
  Interventions: Radiation: [11C]PHNO; Drug: Aripiprazole

INTERVENTIONS:
Radiation: [11C]PHNO — examine the effects of [11C]PHNO mass carry-over and displaceable binding
Drug: Aripiprazole — A 4th scan will follow a 15mg dose of aripiprazole (a D2/D3 compound which allows the highest clinically acceptable blockade of central D2/D3 receptors)

SUMMARY:
This will be an open label, non-randomised [11C]PHNO PET study using healthy male volunteers. Each volunteer will undergo 4 [11C]PHNO PET scans to allow for further characterisation of this radioligand and examine the effects of [11C]PHNO mass carry-over and displaceable binding in the brain. This study aims to obtain data from 6 evaluable subjects.

DETAILED DESCRIPTION:
A test-retest (TRT) investigation of [11C]PHNO in human is required to further characterise [11C]PHNO. [11C] PHNO possesses very high affinity for the D3 receptor, and therefore most clinical studies are conducted at D3 occupancies >10%. As [11C]PHNO kinetics in the target brain regions are moderately slow, considerable mass carry over may be present on a 2nd PET scan conducted on the same day. In addition there appears to be a significant displaceable binding component in the cerebellum, which, if not accounted for, will lead to a bias in the quantification of specific [11C]PHNO binding. The aim of this study is therefore to examine the effects of [11C]PHNO mass carry-over and displaceable binding in the cerebellum, on the quantification of [11C]PHNO PET data.

This will be an open label, non-randomised [11C]PHNO PET study using healthy volunteers. Each volunteer will undergo 4 [11C]PHNO PET scans:

1st and 2nd scans; TRT on the same day with a minimal gap between [11C]PHNO injections to examine the effects of PHNO mass carry over, 3rd scan >1 week later to determine the "true" TRT variability and a 4th scan will follow a 15mg dose of aripiprazole (a D2/D3 compound which allows the highest clinically acceptable blockade of central D2/D3 receptors) and will examine the amount of displaceable binding in the cerebellum, a proposed reference tissue for [11C]PHNO.

The scan data will be quantified as regional volumes of distribution (VT).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible physician
2. Male subjects between 25 and 55 years of age.
3. Male subjects must agree to use one of the contraception methods listed
4. Capable of giving written informed consent

Exclusion Criteria:

1. The subject has a positive pre-study drug/alcohol screen
2. The subjects is using or has used regular prescription or non-prescription drugs
3. Current or recent (within one year) gastrointestinal disease
4. A screening ECG with a QTc value of >450msec and/or a PR interval outside the range 120 to 200msec or an ECG that is not suitable for QT measurements
5. Pulse rate <50 or >100 bpm OR a systolic blood pressure >140 or <100 OR a diastolic blood pressure >90 or <60.
6. History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
7. Any previous or current psychiatric diagnosis listed in DSM-IV Axis I or II
8. Any history of suicidal attempts, suicidal ideation or behaviour as assessed by appropriately trained study personnel.
9. History of alcohol dependence
10. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
11. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
12. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
13. Where participation in the study would result in donation of blood or blood products in excess of 550 mL within a 56 day period.
14. Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden
15. Family history of cancer
16. History of claustrophobia or subjects feeling that he will be unable to lie still on his back in the PET camera for a period of ~2 hours at a time.
17. History or presence of a neurological diagnosis
18. Presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies as assessed by a standard pre-MRI questionnaire.
19. Unwillingness or inability to follow the procedures outlined in the protocol. -

Ages: 22 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
volume of distribution | one year
  Regional volume of distribution (VT) in sub-cortical, brainstem and cerebellar regions of interest at each PET scan.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, London, United Kingdom